CLINICAL TRIAL: NCT04179981
Title: Impact of Positive Airway Pressure Therapy on Clinical Outcomes in Older Veterans With Chronic Obstructive Pulmonary Disease and Comorbid Obstructive Sleep Apnea (Overlap Syndrome)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E3124-R
Record Dates: First submitted 2019-11-25; First posted 2019-11-27 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Sleep Apnea Syndrome; Obstructive Sleep Apnea; COPD; Overlap Syndrome; Quality of Life; Neurocognitive Function; Sleepiness; Elderly; Positive Airway Pressure
Keywords: Apnea; Sleep Apnea Syndromes; Sleep Apnea, Obstructive; Nervous System Diseases; Respiration Disorders; Respiratory Tract Diseases; Signs and Symptoms, Respiratory; positive airway pressure; cognitive function; quality of life; sleepiness
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Obstructive; Pulmonary Disease, Chronic Obstructive; Sleepiness; Apnea; Nervous System Diseases; Respiration Disorders; Respiratory Tract Diseases; Signs and Symptoms, Respiratory

STUDY DESIGN:
Intervention Model Description: Comparing outcomes in patients with OVS after randomization to PAP therapy vs. conservative care in a parallel group fashion
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Conservative care (control arm) (Other): Eligible OVS patients will receive conservative care/usual care with education about sleep apnea and sleep hygiene via handouts and video instructions. This is the control arm.
  Interventions: Other: Conservative care (control arm)
- PAP therapy arm (Active Comparator): PAP Therapy will be provided to eligible patients with OVS. This is the active therapy arm.
  Interventions: Device: Positive airway pressure

INTERVENTIONS:
Device: Positive airway pressure — Positive airway pressure therapy. OVS patients randomized to PAP therapy arm will be titrated to optimal PAP therapy per standard protocol and assigned to use PAP therapy.
  Arms: PAP therapy arm
Other: Conservative care (control arm) — Eligible OVS patients will receive conservative care/usual care with education about sleep apnea and sleep hygiene via handouts and video instructions. This is the control arm.
  Arms: Conservative care (control arm)

SUMMARY:
Obstructive sleep apnea (OSA) and Chronic Obstructive Pulmonary Disease (COPD) are highly prevalent chronic respiratory diseases in the Veteran population. OSA co-occurring with COPD, known as Overlap Syndrome (OVS), is a complex chronic medical condition associated with grave consequences. OVS is highly prevalent in Veterans. Veterans with OVS may be at increased risk for cognitive deficits, poor sleep quality as well as a reduced quality of life (QoL). The overall objective is to study the effects of positive airway pressure therapy on clinical outcomes in patients with OVS.

DETAILED DESCRIPTION:
There are no studies regarding the impact of PAP therapy on sleep disturbance, cognitive function and quality of life in patients with OVS. The investigators' rationale is that in patients with moderate-severe OVS, PAP therapy will effectively alleviate sleepiness, sleep disturbances and cognitive deficits, and, thereby, improve QoL. 'PAP' includes either continuous positive airway pressure (CPAP) or noninvasive positive airway pressure ventilation (NIPPV).

Objectives:

Specifically, the investigators will study the effectiveness of PAP therapy vs. conservative care in reducing daytime sleepiness and in improving sleep quality and QoL in older Veterans with OVS.

The investigators will also explore whether CPAP is non-inferior to noninvasive positive airway pressure ventilation (NIPPV) in reducing daytime sleepiness, sleep disturbances and neurocognitive dysfunction, and in improving QoL in older Veterans with OVS.

ELIGIBILITY:
Inclusion Criteria:

* OSA with moderate-to-severe disease, AHI 20 per hour by in-lab polysomnography with concomitant moderate-severe COPD based on pulmonary function tests (PFTS) and with past significant history (>10 pack-years) of smoking
* Male or female gender
* Age greater than or equal to 60 years
* Stable treatment regimen for COPD

Exclusion Criteria:

* Current or prior treatment with PAP or oral appliance
* Central sleep apnea defined as central apnea index >5 per hour and comprising 50% of AHI
* Known primary neuromuscular diseases
* Disorders that may impact cognitive function including:

  * neurodegenerative disorders
  * traumatic brain injury
* untreated PTSD and/or history of learning disability
* Medicines that may cause or alter sleepiness: sedative hypnotics, or stimulants as these may alter the results
* Patient is actively suicidal due to depression, unstable mental health condition
* Epworth sleepiness score >16 (severe sleepiness) or a near-miss or prior automobile accident due to sleepiness within the past 12 months
* Narcolepsy is the primary sleep disorder, with requirement of stimulant medications
* Employed as a commercial driver or operating heavy machinery
* On long-term oxygen therapy prior to start of study, more than 12 hr/day
* Patients is unable to use either a nasal or face mask (e.g., facial trauma, claustrophobia)
* Consumption of >3 alcoholic beverages per day or current use of some illicit drugs, as these may contribute to cognitive deficits
* Patients who cannot give informed consent
* Patients receiving hospice care
* Pregnant women due to unknown risks

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 668 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Neurocognitive function Trails A and Trails B | Change from baseline at 3 and 6 months
  Trails A and Trails B test will be administered to evaluate attention and psychomotor function. This score is adjusted for age, race, gender, and years of education. Scored on a Standard scale of 100 +/- 15 for normal ranges, above 115 is above average, below 85 is considered below average.
Neurocognitive function PASAT | Change from baseline at 3 and 6 months
  PASAT (Paced Auditory Serial Addition Test) will be administered to evaluate vigilance and executive function. The PASAT is recorded as the total number of correct responses (from 0-60), or the percent of correct responses out of 60 (from 0-100), where a higher value is a better outcome.
Neurocognitive function Stroop color-word interference | Change from baseline at 3 and 6 months
  Stroop color-word interference test will be administered to evaluate executive function. This score is adjusted for age, and years of education. Scored on a Standard scale of 100 +/- 15 for normal ranges, above 115 is above average, below 85 is considered below average.
Neurocognitive function DIGIT | Change from baseline at 3 and 6 months
  DIGIT test will be administered to evaluate short-term and working memory. This score is adjusted for age. Scored on a Standard scale of 100 +/- 15 for normal ranges, above 115 is above average, below 85 is considered below average.
Neurocognitive function WASI | Change from baseline at 3 and 6 months
  Abbreviated Wechsler Abbreviated Scale of Intelligence (WASI) will be administered to evaluate verbal comprehension and working memory. This score is adjusted for age. Scored on a Standard scale of 100 +/- 15 for normal ranges, above 115 is above average, below 85 is considered below average.
Neurocognitive function WMS | Change from baseline at 3 and 6 months
  Wechsler Memory test (WMS) will be administered to measure Verbal comprehension, and working and visual memory. Scored on a Standard scale of 100 +/- 15, where a higher score is a better outcome.
Neurocognitive function PVT | Change from baseline at 3 and 6 months
  Psychomotor Vigilance Test (PVT) will be administered to measure Alertness and vigilance, in terms of number of lapses and reaction time. The performance score ranges from 0-100, where a higher value is a better outcome.
Neurocognitive function HVLT-R | Change from baseline at 3 and 6 months
  Hopkins Verbal Learning Test - Revised (HVLT-R) will be administered to evaluate Verbal learning and memory. Scored on a Standard scale of 100 +/- 15, where a higher score is a better outcome.
Sleepiness ESS | Change from baseline at 3 and 6 months
  Epworth sleepiness scale (ESS) score will be measured. This score is on a scale of 0-24, where a higher value indicates greater degree of sleepiness.
Sleep quality PSQI | Change from baseline at 3 and 6 months
  Pittsburgh Sleep Quality Index (PSQI) is a detailed assessment of subject sleep quality over the most recent month by considering seven "component" scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The sum of scores for these seven components yields one global score to assess sleep quality on a scale of "poor" to "good".
Quality of life SF-36v2 | Change from baseline at 3 and 6 months
  QoL will be assessed using the survey SF-36v2 Health survey. Thirty-five of the SF-36v2 items are used to measure eight domains of health-related quality of life. These are on a scale of 0-100, where higher values indicate a better outcome.
Quality of life FOSQ | Change from baseline at 3 and 6 months
  Disease specific QoL will be assessed using the Functional Outcomes of Sleep Questionnaire FOSQ/(FOSQ). There are 5 subscale domains of the FOSQ (General Productivity, Social Outcome, Activity Level, Vigilance, and Intimate Relationships and Sexual Activity). There all range from 0-20, where a higher value is a better outcome. The total FOSQ is the sum of these subscale domains and ranges from 0-100, where a higher value is a better outcome.
Quality of life SGRQ | Change from baseline at 3 and 6 months
  Disease specific QoL will be assessed using the St. George's Respiratory Questionnaire (SGRQ). The SGRQ has three subscale domains (Symptoms, Activity, and Impacts), which range from 0-100, where a higher value indicates a worse outcome. The total SGRQ is the average of these subscale domains and is on a scale of 0-100, where a higher value is a worse outcome.

SECONDARY OUTCOMES:
Hours of nightly positive airway pressure (PAP) use | Change from baseline at 3 and 6 months
  Collection of PAP adherence data from the smart card of the PAP machine or from online data.
Patient preferance for type of PAP (PAP arm) | at 3 and 6 months
  A visual analog scale to determine preference to CPAP vs NIPPV therapy. A scores will range from -10 to +10, where a higher score is better.
Fatigue severity | Change from baseline at 3 and 6 months
  Fatigue Severity Scale (FSS): FSS measures how fatigue affects motivation, exercise, physical functioning, carrying out duties, interfering with work, family, or social life. Where a higher value is a worse outcome.
Sleep-dependent memory | At baseline and at 3 months
  In a subgroup of patients, the investigators will perform Word-pair test and PVT before and after sleep period, this is an exploratory measure.
Blood CO2 or bicarbonate level | At baseline and at 6 months
  Test is being done to evaluate for presence or absence of hypercapnia

CONTACTS AND LOCATIONS:
Overall Officials: Susmita Chowdhuri, MD MS, Principal Investigator — John D. Dingell VA Medical Center, Detroit, MI
Locations (1):
- John D. Dingell VA Medical Center, Detroit, MI, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No